CLINICAL TRIAL: NCT03958409
Title: Evaluation and Management of Metabolic Bone Disease in Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2000022066
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Skeletal Anomalies; Kidney Transplant; Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rigorous evaluation (Experimental): Participants will be evaluated for the rigorous evaluation received.
  Interventions: Diagnostic Test: measurements to evaluate metabolic bone disease
- Standard care (Active Comparator): The participants will be evaluated for the standard of care received.
  Interventions: Diagnostic Test: standard care

INTERVENTIONS:
Diagnostic Test: measurements to evaluate metabolic bone disease — The participants will be evaluated for a) Mineral metabolism: blood calcium, phosphorus, PTH, 25(OH) vitamin D; b) Bone turnover markers: bone-specific alkaline phosphatase, cross-linked C-telopeptide of type I collagen (CTx), and N-terminal propeptide of type I collagen (PINP); c) Bone Mineral Density using a Dual energy x-ray absorptiometry which is the standard method by which bone mass is measured clinically. The bone mass at the lumbar spine, wrist, hip and total body bone mass at 3, and 18 months.
  Arms: Rigorous evaluation
Diagnostic Test: standard care — Blood tests (Ca, Phos, PTH- mineral lab, 25OHVitD);Pregnancy Test (if applicable); dual energy X-ray absorptiometry (DXA); Bone Biopsy only if clinically indicated; treatment as clinically indicated.
  Arms: Standard care

SUMMARY:
There is a well-documented increased risk for disordered mineral bone homeostasis in Kidney Transplant Recipients (KTRs) when compared to the general population, leading to a markedly increased risk for fragility fractures and their associated morbidity and mortality. A more uniform and rigorous evaluation of bone and mineral homeostasis,than is afforded to patients under "normal care", will result in better clinical outcomes in KTRs.

DETAILED DESCRIPTION:
The aim is to comprehensively characterize the mineral metabolism and skeletal phenotype in kidney transplant recipients (KTRs) to being to identify risk factors for post-kidney transplant mineral bone disease (PKT-MBD); and to evaluate whether treatment of abnormalities in these parameters will improve skeletal health as quantified by bone mineral density (BMD), bone turnover markers (rate of skeletal remodeling) and Osteoprobe (a direct index of bone quality using reference point indentation technology.

Participants in the rigorous evaluation arm will be followed with a) Mineral metabolism: blood calcium, phosphorus, parathyroid hormone (PTH), 25(OH) vitamin D; b) Bone turnover markers: bone-specific alkaline phosphatase, cross-linked C-telopeptide of type I collagen (CTx), and N-terminal propeptide of type I collagen (PINP); c)Bone Mineral Density using a Dual energy x-ray absorptiometry which is the standard method by which bone mass is measured clinically.

NOTE: The use of the Osteoprobe was discontinued on 9/5/19 due to safety concerns from the FDA about the device in other trials/other sites.

The Control Cohort is essentially an historical control group who will have received standard of care for the 18 months ending just prior to the enrollment of our Intervention Cohort. A coincident Control Cohort will not be used because knowledge of the additional data to be collected in the Control Cohort will undoubtedly influence their care by their attending nephrologists and surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant subjects within the first 3 months after surgery (intervention cohort) and 18 months after surgery (control cohort)
* Age between 30 to 65 years old
* Estimated glomerular filtration rate (GFR) > 35 ml/min/1.73 m2

Exclusion Criteria:

* Major acute post-operatory complications (infection, urine leak, delayed graft function)
* Living related-donor KTRs
* Estimated GFR ≤ 35 ml/min/1.73 m2
* Significant skin disorder, bruising, local edema, skin infection or are being treated with anticoagulants (such as warfarin, heparin, low molecular weight heparin or direct thrombin inhibitors) or have known or acquired clotting disorders since the OsteoProbe® procedure would be unsafe
* Patients who do not plan to be followed at Yale New Haven for at least 18 months
* Morbidly obese (BMI >40)
* History of gastroparesis

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Change in bone turnover marker carboxy-terminal collagen crosslinks (CTx) | 18 months
  In the intervention group changes in measures of mineral metabolism (serum calcium, phosphorus, PTH and 25 OH vitamin D levels), changes in bone turnover markers, BMD and bone quality markers will be compared to baseline results. The primary outcome variable will be the change in serum CTx from baseline. CTx is a marker of bone resorption and rates of resorption predict bone loss and fracture risk.

SECONDARY OUTCOMES:
Variance in bone loss | 18 months
  the changes in PTH, CTx, Procollagen Type 1 N-Terminal Propeptide (P1NP), Trabecular Bone Score (TBS) and Bone Material Strength Index (BMSi) will be correlated with changes in bone mineral density (BMD) in a multiple regression model to determine their contributions to the variance in rates of bone loss. This will serve to inform our planned prospective study in terms of what measures to follow.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Belfort de Aguiar, Phd,MD, Principal Investigator — Yale University
Locations (1):
- Yale Transplantation Center/Yale-New Haven Hospital, New Haven, Connecticut, United States